CLINICAL TRIAL: NCT01911325
Title: A Phase Ib/II Study of Docetaxel With or Without Buparlisib as Second Line Therapy for Patients With Advanced or Metastatic Squamous Non-small Cell Lung Cancer
Brief Title: Phase II Study of Buparlisib + Docetaxel in Advanced or Metastatic Squamous Non-small Cell Lung Cancer (NSCLC) Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Review of safety and preliminary efficacy data showed marginal anti-tumor activity.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBKM120D2205; 2013-000833-11 (EudraCT Number)
Record Dates: First submitted 2013-05-16; First posted 2013-07-30 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Squamous Non-small Cell Lung Cancer
Keywords: Squamous non-small cell lung cancer; NSCLC; Docetaxel; Buparlisib; BKM120; Metastatic; Stage IIIb; Stage IV; PI3K inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — NVP-BKM120; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase Ib: Buparlisib + docetaxel (Experimental): Buparlisib (BKM120) oral once daily: 80 mg and 100 mg dose levels to be tested in the dose escalation part of the trial in combination with docetaxel every three week intravenous (i.v.) infusion: 75 mg/m2 as per label.
  Interventions: Drug: Buparlisib; Drug: Docetaxel
- Phase II: Buparlisib + docetaxel (Experimental): Buparlisib oral once daily: MTD/RP2D mg to be tested in combination with docetaxel every three week i.v. infusion: 75 mg/m2 as per label.
  Interventions: Drug: Buparlisib; Drug: Docetaxel
- Phase II: Placebo + docetaxel (Placebo Comparator): Buparlisib matching placebo oral once daily to be tested in combination with docetaxel every three week i.v. infusion: 75 mg/m2 as per label.
  Interventions: Drug: Buparlisib matching placebo; Drug: Docetaxel

INTERVENTIONS:
Drug: Buparlisib
  Other Names: BKM120
  Arms: Phase II: Buparlisib + docetaxel; Phase Ib: Buparlisib + docetaxel
Drug: Buparlisib matching placebo
  Arms: Phase II: Placebo + docetaxel
Drug: Docetaxel

SUMMARY:
This is a multi-center, open-label Phase Ib dose escalation part followed by a randomized double-blinded placebo controlled Phase II part.

The Phase Ib part will determine the Maximum Tolerated Dose (MTD)/Recommended Phase II Dose (RP2D) of buparlisib in combination with docetaxel. Subsequently the MTD/RP2D will be investigated in a Phase II randomized trial in patients with advanced or metastatic squamous NSCLC.

DETAILED DESCRIPTION:
Based on an overall review of safety and preliminary efficacy data done on 01-Dec-2014 showing marginal anti-tumor activity and newly emerged treatment options, a decision was taken to stop further development of this combination in patients with advanced or metastatic squamous NSCLC and Phase II of the study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult ≥ 18 years old at the time of informed consent
* Patient has histologically and/or cytologically confirmed diagnosis of squamous NSCLC. Diagnosis of mixed squamous and non-squamous or adenosquamous NSCLC will be acceptable for enrollment.
* Patient has received one prior approved regimen of platinum-based chemotherapy (excluding a docetaxel-containing regimen) for advanced or metastatic (Stage IIIb or Stage IV) squamous NSCLC, followed by disease progression. A drug provided as maintenance therapy following cytotoxic chemotherapy will be considered to be part of that regimen.

Note: Patients who received paclitaxel therapy are eligible for this trial. •Patient has adequate tumor tissue (either archival or new tumor biopsy) for the analysis of PI3K-related biomarkers.

Enrollment in the Phase II part of the study is contingent on the central laboratory confirming receipt of an adequate amount of tissue including sufficient DNA for analysis.

•Patient has measurable or non-measurable disease according to RECIST version 1.1 criteria.

Phase II only: Patient must have at least one measurable lesion as per RECIST criteria.

* Patient has an ECOG performance status ≤ 1
* Patient has adequate bone marrow and organ function

Exclusion Criteria:

* Patient has received previous treatment with a PI3K or AKT inhibitor
* Patient has symptomatic Central Nervous System (CNS) metastases Patients with asymptomatic CNS metastases may participate in this trial. The patient must have completed prior local treatment, if any, for CNS metastases ≥ 28 days prior to the start of study treatment (including radiotherapy and/or surgery, or ≥ 14 days for stereotactic radiosurgery).
* Patient has a score ≥ 12 on the PHQ-9 questionnaire.
* Patient selects a response of "1, 2 or 3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9).
* Patient has a GAD-7 mood scale score ≥ 15.
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation or patients with active severe personality disorders.
* Patient has ≥ CTCAE grade 3 anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Incidence of Dose Limiting Toxicities (DLTs) in Cycle 1 | Day 21
  To determine the maximum tolerated dose/recommended phase ll dose (MTD/RP2D) of buparlisib in combination with docetaxel by assessing the incidence of DLTs in Cycle 1; Cycle 1 = 21 days
Phase II: Progression Free Survival (PFS) | After 70 PFS events have been observed at 9 months after patient enrollment
  PFS as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. To estimate the treatment effect of docetaxel and buparlisib or placebo on PFS in patients with advanced or metastatic squamous NSCLC.

SECONDARY OUTCOMES:
Number of patients with at least one adverse event. | Up to 30 days after the last dose
Number of patients with laboratory abnormalities. | Up to 30 days after the last dose
Overall Survival (OS) | Treatment start (phase Ib)/randomization (phase II), every 6 weeks to the date of first document progression for up to 3 years
  Overall survival (OS) time is measured from the start of study drug to the date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact. Data will be collected post treatment every 6 weeks until approximately 75% of patients have reached the survival endpoint (Phase I + Phase II)
Overall response rate (ORR) | Every 6 weeks from randomization until first documented progression for up to 3 years
  Overall response is the number of participants who had a complete response (CR) or a partial response (PR) based on local investigator's assessment of RECIST 1.1 criteria.
Time to response (ToR) | Every 6 weeks from randomization until first documented progression for up to 3 years
  Time to overall response is defined as the time from the date of first drug intake in Phase Ib and from the date of randomization in Phase II to the date of first documented response.
Duration of response (DR) | Every 6 weeks from randomization until first documented progression for up to 3 years
  Duration of overall response is defined as the elapsed time between the date of first documented response and the following date of event defined as the first documented progression or death due to underlying cancer.
Change in electrocardiogram (ECG) and cardiac imaging | Up to 30 days after the last dose
Changes in vital signs | Up to 30 days after the last dose
Shift in ECOG performance status | Baseline, worst post-baseline result at day 1 of every cycle and at end of study treatment (3 years)
  cycle = 21 days; end of treatment is defined as 15 days after treatment discontinuation; There is no treatment duration as patients continue to receive drug till toxicity or they withdraw consent
Change in Mood scales | Up to 30 days after the last dose
Time to definitive 10% deterioration in the global health status/quality of life (QOL) scale score of the EORTC QLQ-C30 | Baseline, Every 6 weeks until disease progression for up to 3 years
  Date of event is defined as at least 10% relative to baseline worsening of the corresponding scale score or death due to any cause
Change in the global health status/quality of life (QOL) scale score of the EORTC QLQ-C30 | Baseline, Every 6 weeks until disease progression for up to 3 years
  Change in the domain scores
Docetaxel and buparlisib plasma concentrations | Cycle 1 day 8 and 15, Cycle 2-Cycle n day 1
PFS Phase Ib | at 3 months after patient enrollment, every 6 weeks until disease progression for up to 3 years
  PFS as per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (4):
  - Highlands Oncology Group SC-1, Fayetteville, Arkansas
  - H. Lee Moffitt Cancer Center & Research Institute H Lee Moffitt, Tampa, Florida
  - Reliant Medical Group Reliant Medical Group, Worcester, Massachusetts
  - Virginia Oncology Associates Virginia Oncology Assoc. (2), Norfolk, Virginia
- Belgium (2):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Mons
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Saint-Herblain
- Germany (3):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Monza, MB, Italy
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Stockholm, Sweden